CLINICAL TRIAL: NCT03704025
Title: Effects of Virtual Physiotherapy on Exercise Training in Cardiac Patients
Brief Title: Home-based Exercise Training in Cardiac Patients
Acronym: VAPA-Oulu
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Business Finland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 281/2016
Record Dates: First submitted 2018-06-01; First posted 2018-10-12 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Physical Fitness; Patient Adherence; Quality of Life; Autonomic Nervous System Imbalance
Keywords: Exercise tolerance; Heart rate variability; Baroreflex sensitivity
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Current guidelines rehabilitation (Active Comparator): Exercise rehabilitation at home according to current guidelines. Training is guided and controlled by diary.
  Interventions: Behavioral: Current guidelines rehabilitation
- Mobile device guided rehabilitation (Experimental): Exercise rehabilitation at home according to current guidelines. Training is guided and controlled by virtual augmented reality glasses or by mobile device.
  Interventions: Behavioral: Mobile device guided rehabilitation

INTERVENTIONS:
Behavioral: Current guidelines rehabilitation — Exercise training intervention is six months and includes four to five aerobic and two strength training session a week according to American Heart Association guidelines for coronary artery disease patients. All the patients will have a detailed and personalized training diary.
  Arms: Current guidelines rehabilitation
Behavioral: Mobile device guided rehabilitation — Exercise training intervention is six months and includes four to five aerobic and two strength training session a week according to American Heart Association guidelines for coronary artery disease patients. Study group will have virtual glasses or mobile device to motivate and control exercise training program.
  Arms: Mobile device guided rehabilitation

SUMMARY:
The investigators hypothesize that exercise training program guided by virtual augmented reality glasses or by video from computer screen used at home will improve motivation into exercise training and results in superior adherence to exercise training compared to current practice. The primary objectives of this research project are to study the effects of exercise training guidance by novel technology on 1) exercise capacity, 2) adherence to exercise training, 3) changes in cardiac autonomic function and 4) quality of life in acute coronary syndrome (ACS) patients.

DETAILED DESCRIPTION:
The subjects of the study will be recruited from the consecutive series of patients of men and women admitted to Oulu University Hospital due to an acute coronary syndrome (ACS). The study population will be randomized into control group (n=25) and study group (n=25) matched with age and gender. For all subjects, clinical status including quality of life questionnaire, exercise capacity and autonomic function measurements will be performed at baseline and after exercise training. Exercise training program is six months for both groups according to current guidelines. All the patients will have a detailed and personalized training prescription. Study group will have virtual augmented reality glasses or computer with training video to motivate and control exercise training prescription at home.

ELIGIBILITY:
Inclusion Criteria:

* Recent (< 1 month) acute coronary syndrome

Exclusion Criteria:

* New York Heart Association (NYHA) functional classification class IV (heart failure)
* unstable chest pain (angina pectoris, Canadian Cardiovascular Society grading of angina pectoris class 4)
* ST-segment elevation myocardial infarction (STEMI)
* implanted cardioverter defibrillation or pacemaker (or planned)
* chronic atrial fibrillation
* musculoskeletal disorder (unable to participate exercise training)
* participation in competing clinical trial
* severe peripheral atherosclerosis
* retinopathy or neuropathy
* dementia
* life-expectancy due to other serious disease < 2 years or any other reason why patient is unable or unwilling to provide written informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-01-05 (Actual)

PRIMARY OUTCOMES:
Change in exercise capacity | Six months (baseline and 6 months)
  Change in maximal load during exercise stress test (metabolic equivalents)

SECONDARY OUTCOMES:
Adherence to exercise rehabilitation | Weekly from baseline to six months
  Realized training in relation to prescribed training over six months
Change in the standard deviation of normal to normal intervals (SDNN) of heart rate variability | Six months (baseline and 6 months)
  Change in 24 h SDNN (ms)
Change in very low frequency (VLF) of heart rate variability | Six months (baseline and 6 months)
  Change in 24 h VLF (ms^2)
Change in low frequency (LF) of heart rate variability | Six months (baseline and 6 months)
  Change in 24 h LF (ms^2)
Change in high frequency (HF) of heart rate variability | Six months (baseline and 6 months)
  Change in 24 h HF (ms^2)
Change in fractal scaling exponent of heart rate variability | Six months (baseline and 6 months)
  Change in 24 h Fractal scaling exponent (a.u.)
Change in baroreflex sensitivity | Six months (baseline and 6 months)
  Change in spontaneous baroreflex sensitivity by cross-spectral method (ms/mmHg)
Change in quality of life | Six months (baseline and 6 months)
  Change in quality of life measured by 15-D questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Mikko P Tulppo, PhD, Principal Investigator — University of Oulu
Locations (1):
- University of Oulu, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saarikoski EO, Roiha ETM, Kiviniemi AM, Cerdan-De-Las-Heras J, Perkiomaki J, Kaikkonen KS, Tulppo MP. Adherence to exercise after an acute coronary syndrome: a 6-month randomized controlled trial. Front Physiol. 2024 Jan 26;15:1319907. doi: 10.3389/fphys.2024.1319907. eCollection 2024. PMID 38343424
- [Derived] Dibben G, Faulkner J, Oldridge N, Rees K, Thompson DR, Zwisler AD, Taylor RS. Exercise-based cardiac rehabilitation for coronary heart disease. Cochrane Database Syst Rev. 2021 Nov 6;11(11):CD001800. doi: 10.1002/14651858.CD001800.pub4. PMID 34741536